CLINICAL TRIAL: NCT04759963
Title: Impact of Obstetric Epidural Anesthesia on Mechanical Function of Low Back
Brief Title: Impact of Epidural Anesthesia on Low Back Function
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Assistant Lecturer, South Valley University
Other Study IDs: South Valley University
Record Dates: First submitted 2021-01-23; First posted 2021-02-18 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: follow up for 6 women who gave birth through a cesarean delivery with Midline approach epidural anesthesia. They will perform all assessment procedures: Visual analog scale (VAS) and Oswestry Disability Index (ODI).
- Group B: follow up for 13 women who gave birth through a cesarean delivery with Midline approach spinal anesthesia. They will perform all assessment procedures: Visual analog scale (VAS) and Oswestry Disability Index (ODI).
- Group C: follow up for 7 women who gave birth through a cesarean delivery with general anesthesia. They will perform all assessment procedures: Visual analog scale (VAS) and Oswestry Disability Index (ODI).
- Group D: follow up for 12 women who are the control group (who did not experience any pregnancy or anesthesia. They will perform all assessment procedures: Visual analog scale (VAS) and Oswestry Disability Index (ODI).

SUMMARY:
Back pain is a common complication after the use of epidural anesthesia in obstetric and non-obstetric surgeries and occurs in 30-45% of cases (Brown, 2005). Certain psychological problems such as depression or unhappiness due to loss of employment may prolong the episode of low back pain (Miller, 2012). According to Egyptian Institution of Health Metrics and Evaluation (IHME), Low Back Pain is the first cause of disability in Egypt from 2007 to 2017.

So, this study will investigate if midline approach of obstetric epidural anaesthesia will be a relative risk for subacute low back mechanical functions as a new way to examine if this type of anaesthesia is involved in the presence of subacute negative effects on the mechanical function of low back or not (to resolve the controversy).

DETAILED DESCRIPTION:
The lumbar (or lower back) region is made up of five vertebrae (L1-L5), sometimes including the sacrum. Stability of the spine is provided by the ligaments and muscles of the back and abdomen (Floyd and Thompson, 2008).

The primary biomechanical function of the spine is to provide structural support, to allow the body to move freely, and to protect the spinal cord and nerves. Muscles balance external loads to the spine, which supports the load and allows for the motion through its multilevel joint arrangement (Dreischarf et al., 2016).

Low back pain (LBP) is a common minor yet unpleasant complication after epidural anesthesia. Different mechanisms are suggested such as needle trauma and myotoxicity of local anesthetic (Louizos et al., 2005) and incidence of backache after epidural anaesthesia might be expected to be higher than that after spinal anaesthesia (Brown and Elman, 1961).

In most episodes of low back pain, a specific underlying cause is not identified or even looked for, with the pain believed to be due to mechanical problems such as muscle or joint strain (Casazza, 2012). Most cases are idiopathic but usually attributable to muscle strain or ligament injury; found in 65% to 70% of patients with mechanical chronic back pain (Cohen et al., 2008) while totally mechanical low back pain is reported as the cause in about 80% to 95% of patients with low back pain (Cohen et al., 2008) & (Dixit, 2017).

Caesarean section is when a baby is born through an incision in the mother's abdomen and uterine wall. This requires effective anaesthesia which can be regional (epidural or spinal) or a general anaesthetic. With regional epidural anaesthesia, the anaesthetic is infused into the space around the mother's spinal column, whilst with regional spinal anaesthesia, the drug is injected as a single dose into the mother's spinal column. With the two types of regional anaesthesia, the mother is awake for the birth but numbed from the waist down while with general anaesthesia, the mother is unconscious for the birth with the anaesthetic affecting her whole body (Afolabi and Lesi, 2012).

The epidural needle can be placed using the midline or paramedian approach. In both cases, lidocaine 1% is infiltrated in the epidural needle insertion area.

In the midline approach technique, the needle is placed in the midline between 2 spine processes. In the paramedian approach technique, the needle is inserted 1 cm lateral and 1 cm caudal to the lower border of the upper spinous process.

The epidural needle in the medline approach is advanced through ligaments: supraspinous ligament, interspinous ligament, ligamentum flavum and into the target epidural space. Each ligament has different density and texture, which affects the feel of the needle and the resistance to insertion (Vaughan et al., 2013).

Some explanations for Low Back Dysfunction after Epidural Anaesthesia:

The incidence of back pain after epidural anesthesia is over 20% (Rose, 2012) & (Saghafinia et al., 2009) & (Muslu et al., 2009). It occurs rarely after spinal anesthesia (Schwabe and Hopf, 2001). This indicates that back pain may be associated with local trauma and nerve injury caused by the epidural needle, leading to aseptic periosteitis, tendonitis, ligamentous inflammation and/or osteochondritis, which result in lumbar pain (Kalso, 2013).

* Excessive elongation of spinal ligaments can cause micro-trauma of the ligament fibers and tears or ruptures occur. Also, the interspinous ligaments are the first structures damaged (excessive stretching) when the spine is hyperflexed (Adams et al., 1998).
* Degeneration and excessive stress on the thoracolumbar fascia may also cause micro-trauma, and resulting in tears. Thoracolumbar fascia may become damaged by over-stretching or excessive stress, potentially eliciting pain (Bogduk, 1983).
* Other contributing factors include needle trauma, surgical positioning, injection of saline or local anesthetic into the interspinous ligaments and development of a supraspinous hematoma (Covet et al., 1967), (Crawford, 1972).
* Excessive stretching of ligaments after relaxation of paraspinal muscles and localized trauma to the intervertebral disc has also been implicated in causing back pain (Agarwal and Kishore, 2009).

Visual analogue scale (VAS):

The visual analogue scale is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." (Delgado et al., 2018).

Pressure algometry:

Pressure algometry has been described as a semi-objective method, or subjective measure and Pain Pressure Threshold (PPT) is a quantitative sensory test of tissue sensitivity, and it is defined as the minimal amount of pressure that produces pain, measured via a pressure algometer (Ylinen, 2007).

Inclinometers:

An inclinometer or tilt meter is an instrument for measuring angles of slope (or tilt), elevation or depression of an object or body segment with respect to gravity (Nielsen et al., 2011).

Oswestry Disability Index:

The Oswestry Disability Index (ODI) is a valid, reliable, and responsive condition-specific assessment tool that is suited for use in clinical practice. It is easy to administer and score, objectifies clients' complaints, and monitors effects of therapy (Vianin, 2008).

Isokinetic dynamometry:

The isokinetic dynamometer is a gold standard instrument for measuring muscle strength and is safe, valid, and reliable, based on the use of kinetic parameters that also include the angular measurement of a corporeal segment throughout the range of motion (Gonosova et al., 2018) & (Habets et al., 2018) & (Roth et al., 2017) & (Guilhem et al., 2014).

Ultrasound Elastography:

Ultrasound elastography (EUS) is a recently developed ultrasound-based method, which allows the qualitative visual or quantitative measurements of the mechanical properties of tissue (Hall, 2003), (Garra, 2007) & (Garra, 2011).

Myoton Pro Device:

A MyotonPRO (Myoton AS, Estonia) is a portable hand-held myotonometer that can assess muscle tone and soft tissue stiffness. According to prior research, the MyotonPRO is a reliable quantitative measurement for assessing the mechanical properties of muscles (Pruyn et al., 2016).

The MyotonPRO can differentiate the viscoelastic properties of a trigger point from a non-trigger point. Our findings support the reliability of this myotonometer. This affordable and portable tool can be used to objectively measure viscoelastic properties of trigger points (Roch et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* All women gave birth through a cesarean delivery.
* Their ages will range from 18 to 35 years.
* All participants will have body mass index (BMI) not more than 30.
* All participants will be assessed after 6weeks postnatal.
* All participants will be able to continue all assessment procedures.

Exclusion Criteria:

* Women who delivered through vaginal delivery.
* Women who delivered through cesarean delivery but the used anesthetic technique was the paramedian approach of epidural anesthesia.
* Women who have any non-myofascial low back dysfunctions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Primiparous women or Multiparous who did not receive anaesthesia for at least one year prior to the last delivery.
Study Population: 45 women were enrolled in this study with a 20% rate loss of follow-up (i.e. we need at least 38 participants to complete the study). They were selected from the SVU Teaching Hospitals.
  The Participants were classified into 4 groups: -
  Group (A):
  This group included 6 women. They gave birth through a cesarean delivery using Midline approach epidural anesthesia,
  Group (B):
  This group included 13 women. They gave birth through a cesarean delivery using Midline approach spinal anesthesia
  Group (C):
  This group included 7 women. They gave birth through a cesarean delivery using general anesthesia.
  Group (D):
  This group included 12 women. who are the control group,
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Subacute Low Back Pain intensity | assessment will be done at 6 weeks after the use of anaesthesia during Cesarean section
  Subacute Low Back Pain intensity is assessed by Visual Analogue scale: Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 "no pain" and 10 "worst pain."

OTHER OUTCOMES:
Low Back functional ability | assessment will be done at 6 weeks after the use of anaesthesia during Cesarean section
  Low Back functional ability will be assessed by Oswestry Disability Index: It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. where as grading system is : 0 - 4 No disability
  5 - 14 Mild disability
  15 - 24 Moderate disability
  25 - 34 Severe disability
  35 - 50 Completely disabled

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed GA Ali, Msc, Principal Investigator — South Valley University
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy - SVU, Cairo
  - Faculty of physical therapy, South Valley University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided